CLINICAL TRIAL: NCT03381586
Title: QUILT-1.004: A Single Center, Open-label, Pharmacokinetic Study of Subcutaneous ALT-803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA-ALT-803-03-17
Record Dates: First submitted 2017-12-05; First posted 2017-12-22 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: ALT-803; PK
MeSH Terms: interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 1.0 mg/ml ALT-803
  Interventions: Drug: ALT-803
- Group B (Experimental): 2.0 mg/ml ALT-803
  Interventions: Drug: ALT-803

INTERVENTIONS:
Drug: ALT-803 — Subjects randomized to Group A will receive ALT-803 at a concentration of 1.0 mg/mL and subjects randomized to Group B will receive ALT-803 at a concentration of 2.0 mg/mL. Subjects will receive a single 10 µg/kg subQ dose of ALT-803 on Day 1 of study period 1. After a rest period, subjects will receive a single 20 µg/kg subQ dose of ALT-803 on Day 1 of study period 2.

SUMMARY:
This is a single center, open-label, pharmacokinetic study of ALT-803 administered as a subQ injection to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   1. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of subject care.
   2. Subjects must be willing and able to comply with the scheduled visits, study drug dosing schedule, procedures, laboratory tests, and other requirements of the study.
2. Study Population

   1. Body mass index (BMI) must be within the range of 18 to 28 kg/m2. Subjects must weigh between 50 and 100 kg (inclusive).
   2. Subjects must be in good health as determined by past medical history, complete physical examination, vital signs and laboratory tests at screening.
3. Age and Reproductive Status

   1. Men and women, 18 - 65 years of age.
   2. Female participants of childbearing potential must adhere to using a medically accepted method of birth control up to 28 days prior to screening and agree to continue its use during the study or be surgically sterilized (e.g., hysterectomy or tubal ligation) WOCBP must agree to use effective contraception during the study and for at least 1 month following the last dose of the study drug.
   3. WOCBP must have a negative serum pregnancy test < 14 days prior to first dose of the study drug. Non-childbearing is defined as greater than one year postmenopausal or surgically sterilized.
   4. Male subjects must be willing to use barrier contraception (i.e. condoms and spermicide) from the day of dosing until at least 1 month following the last dose of study drug.

Exclusion Criteria:

1. Medical History and Concurrent Diseases

   1. A past medical history of clinically significant 12 lead EKG abnormalities
   2. Subjects with a history of interstitial lung disease and/or pneumonitis.
   3. HIV-positive.
   4. Significant illness within 2 weeks prior to dosing.
   5. Positive hepatitis C serology or active hepatitis B infection.
   6. Known autoimmune disease requiring active treatment. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 4 weeks or 5 half-lives of registration are excluded.
   7. Psychiatric illness/social situations that would limit compliance with study requirements.
   8. Previous malignancies, unless basal or squamous cell carcinoma of the skin or cervical carcinoma in situ with a complete remission achieved at least 5 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
   9. Loss of ≥ 475 mL blood volume or blood donation transfusion of any blood product within 3 months prior to screening.
   10. Other illness or laboratory abnormality that in the opinion of the Investigator should exclude the subject from participating in this study.
2. Prohibited Treatments and/or Restricted Therapies

   1. Use of any prescription drugs within 4 weeks (hormonal methods of contraception are allowed) or less than 5 half-lives prior to dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within 2 weeks or less than 5 half-lives prior to dosing.
   2. Exposure to any investigational drug or placebo within 3 months of first dose of study drug.
   3. Previous treatment or clinical trial participation with monoclonal antibody therapy.
   4. History of drug or alcohol abuse within 12 months prior to dosing, or those who have a positive urine drug test or breath alcohol test at Screening or Baseline.
   5. Transfusion of blood or any blood product within 3 months prior to screening.
   6. History of using nicotine-containing products or smoking more than 5 cigarettes weekly for at least three months prior to the study through the final evaluation.
3. Allergies and Adverse Drug Reaction

   1. History of severe hypersensitivity reactions to other monoclonal antibodies.
   2. Known history of clinically significant drug allergy at Screening or Baseline
4. Sex and Reproductive Status a. Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35228263/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 1.0 mg/ml ALT-803
  ALT-803: Subjects randomized to Group A will receive ALT-803 at a concentration of 1.0 mg/mL. Subjects will receive a single 10 µg/kg subQ dose of ALT-803 on Day 1 of study period 1. After a rest period, subjects will receive a single 20 µg/kg subQ dose of ALT-803 on Day 1 of study period 2.
- Group B: 2.0 mg/ml ALT-803
  ALT-803: Subjects randomized to Group B will receive ALT-803 at a concentration of 2.0 mg/mL. Subjects will receive a single 10 µg/kg subQ dose of ALT-803 on Day 1 of study period 1. After a rest period, subjects will receive a single 20 µg/kg subQ dose of ALT-803 on Day 1 of study period 2.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 10
Completed | 7 | 7
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (11.3) | 42.5 (11.6) | 44 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Healthy Volunteers [Count of Participants; unit: Participants] | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: PK Profile - Half-life (t½)
Description: The period of time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: Up to 192 hours
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 5
Days
  Period 1 (10 μg/kg) | 1.07 (0.813) | 0.55 (0.095)
  Period 2 (20 μg/kg) | 1.02 (0.758) | 0.68 (0.236)

2. Primary Outcome: PK Profile - Apparent (Extravascular) Volume of Distribution (Vz/F)
Description: Apparent volume of distribution is a ratio of the total amount of drug in the body to the plasma concentration of the drugs such that Vd = amount of drug in body/plasma drug concentration.
Time Frame: Up to 192 hours
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 5
mL/kg
  Period 1 - 10 μg/kg | 13900 (12000) | 5360 (2790)
  Period 2 - 20 μg/kg | 15500 (13000) | 11800 (8170)

3. Primary Outcome: PK Profile - Apparent (Extravascular) Clearance (CL/F)
Description: apparent (extravascular) clearance (CL/F)
Time Frame: Up to 192 hours
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 5
mL/day/kg
  Period 1 - 10 µg/kg | 8650 (5450) | 6610 (2680)
  Period 2 - 20 µg/kg | 10500 (5430) | 11000 (4440)

4. Primary Outcome: PK Profile - Maximum Observed Concentration (Cmax)
Description: maximum observed concentration (Cmax)
Time Frame: Up to 192 hours
Population: In Period 2, 3 participants in each arm dropped off the study. In Group A, the 1 additional participant was excluded from the analysis. Subject 0317-001-0020 samples were Not Calculated for Period 1, but they were calculated for Period 2. Hence, the number of subjects with samples was greater in Period 2 than in Period 1.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
pg/mL
  Period 1 - 10 µg/kg | 1150 (945) | 1080 (902)
  Period 2 - 20 µg/kg: number analyzed (Participants) | 6 | 7
  Period 2 - 20 µg/kg | 1900 (1930) | 1490 (921)

5. Primary Outcome: PK Profile - Time of the Observed Maximum Concentration (Tmax)
Description: time of the observed maximum concentration (Tmax)
Time Frame: Up to 192 hours
Population: as for outcome 4
Measure: Median (Full Range); unit: Days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Days
  Period 1 - 10 µg/kg | 0.167 [0.167 to 2.00] | 0.583 [0.167 to 2.00]
  Period 2 - 20 µg/kg: number analyzed (Participants) | 6 | 7
  Period 2 - 20 µg/kg | 1.00 [0.170 to 1.00] | 0.170 [0.170 to 0.171]

6. Primary Outcome: PK Profile - Area Under the Plasma Concentration Curve From Time 0 Through the Last Measurable Concentration (AUC0-t)
Description: area under the plasma concentration curve from time 0 through the last measurable concentration (AUC0-t)
Time Frame: Up to 192 hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Day*pg/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Day*pg/mL
  Period 1 - 10 µg/kg | 1390 (727) | 1240 (706)
  Period 2 - 20 µg/kg: number analyzed (Participants) | 6 | 7
  Period 2 - 20 µg/kg | 2370 (1410) | 1940 (1040)

7. Primary Outcome: PK Profile - Area Under the Plasma Concentration Curve From Time 0 Extrapolated to Infinite Time (AUC0-inf)
Description: area under the plasma concentration curve from time 0 extrapolated to infinite time (AUC0-inf)
Time Frame: Up to 192 hours
Measure: Mean (Standard Deviation); unit: Day*pg/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 6 | 5
Day*pg/mL
  Period 1 - 10 µg/kg | 1600 (897) | 1740 (731)
  Period 2 - 20 µg/kg | 2420 (1400) | 2130 (1000)

8. Secondary Outcome: Number of Adverse Events
Description: Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Time Frame: Up to 66 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

ADVERSE EVENTS:
Time Frame: Up to 66 days
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=10) | Group B (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1
Myringitis bullous (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Axillary pain (General disorders) | 2 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Chills (General disorders) | 9 | 10
Fatigue (General disorders) | 2 | 0
Feeling of body temperature change (General disorders) | 4 | 8
Injection site reaction (General disorders) | 10 | 10
Malaise (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 7
Fungal skin infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 7
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 1 | 0
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03381586/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03381586/SAP_001.pdf